CLINICAL TRIAL: NCT07059052
Title: Impact of Illness Perception on Quality of Life in Patients With Colorectal Cancer and Ascites
Brief Title: Illness Perception and Quality of Life in Colorectal Cancer With Ascites
Status: Completed | Type: Observational
Sponsor: Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government)
Responsible Party: Principal Investigator, Xujin Guo, Principal Investigator, Hebei Provincial Hospital of Traditional Chinese Medicine
Other Study IDs: 2024021
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer (MSI-H)
Keywords: Illness Perception; Colorectal Cancer with Ascites; Quality of Life; Age; Histological Grade
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Colorectal Cancer and Ascites: A single cohort of 218 patients with a confirmed diagnosis of colorectal cancer and concomitant ascites. These patients were treated at the Hebei Provincial Hospital of Traditional Chinese Medicine between January 2024 and April 2025. Data on their clinical characteristics, illness perceptions, and quality of life were collected at a single point in time for this cross-sectional analysis.

SUMMARY:
This study aimed to investigate the impact of illness perception on the quality of life (QoL) in patients diagnosed with colorectal cancer (CRC) complicated by ascites. The study explores how patients' cognitive and emotional beliefs about their illness relate to their physical, psychological, and social well-being.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a leading cause of cancer-related mortality worldwide, and many patients are diagnosed at advanced stages with complications such as malignant ascites, which severely impairs quality of life (QoL). Illness perception, the framework of beliefs a patient develops about their illness, is known to influence health outcomes. However, this relationship is not well-studied in the specific subgroup of CRC patients with ascites.

This cross-sectional, observational study was designed to fill this gap. A total of 218 patients with CRC and ascites were enrolled. The study collected clinical and demographic data, and assessed illness perception using the Brief Illness Perception Questionnaire (BIPQ) and QoL using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The primary goal was to analyze the correlation between dimensions of illness perception and domains of QoL, and to identify independent clinical and demographic factors that predict patient QoL. The findings are intended to inform the development of targeted psychosocial interventions to improve patient well-being in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of colorectal cancer with ascites, verified by imaging and pathological examination.
* Patient and/or legal guardian provided informed consent.
* Karnofsky Performance Status (KPS) score ≥50.
* Estimated survival ≥6 months.

Exclusion Criteria:

* Presence of other active malignant tumors.
* Severe physical disability precluding participation.
* Severe cardiac, hepatic, or renal dysfunction not related to CRC.
* Presence of severe psychiatric or cognitive disorders.
* History of alcohol or drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included patients diagnosed with colorectal cancer and concomitant ascites. Participants were recruited from those treated at the Hebei Provincial Hospital of Traditional Chinese Medicine between January 2024 and April 2025. All consecutive patients who met the specific inclusion and exclusion criteria during this period and provided informed consent were enrolled in this cross-sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life Score | Assessed once per participant during the study period from January 2024 to April 2025
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30, version 3.0). This 30-item questionnaire evaluates global health status, five functional scales (physical, role, emotional, cognitive, social), and symptom scales. All scores are transformed to a 0-100 scale. For functional scales and global QoL, higher scores represent better functioning or QoL.
Illness Perception Score | Assessed once per participant during the study period from January 2024 to April 2025
  Assessed using the Brief Illness Perception Questionnaire (BIPQ). This 8-item questionnaire evaluates cognitive and emotional representations of illness on a 0-10 scale. The total score ranges from 0 to 80, with higher scores indicating a more threatening or negative illness perception after reverse-scoring relevant items.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Provincial Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei, China